CLINICAL TRIAL: NCT03715907
Title: Financial Incentives for Care Gaps: A Randomized Controlled Trial
Brief Title: Financial Incentives for Care Gaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1805348624
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Delivery of Health Care
Keywords: Professional Practice Gaps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Control: W34 (No Intervention): Members receiving the Control intervention for the W34 (3- to 6-year-old well visit) gap will not receive a mailer.
- Information only: W34 (Experimental): Members receiving the Information Only intervention for the W34 care gap will receive a mailer informing them of that gap, but not of financial incentives for closing the care gap.
  Interventions: Behavioral: Information
- Incentives: W34 (Experimental): Informational W34 mailer and incentive to close gap
  Interventions: Behavioral: Financial Incentives; Behavioral: Information
- Control: LSC (No Intervention): Members receiving the Control intervention for the LSC (lead screening in children) gap will not receive a mailer.
- Information only: LSC (Experimental): Informational LSC mailer and incentive to close gap
  Interventions: Behavioral: Information
- Incentives: LSC (Experimental): Members receiving the Incentives intervention for the LSC care gap will receive a mailer informing them of the gap and eligibility for a gift card if they close the gap.
  Interventions: Behavioral: Financial Incentives; Behavioral: Information
- Control: IMA (No Intervention): No mailer for IMA (immunizations) gap
- Information only: IMA (Experimental): Informational IMA mailer
  Interventions: Behavioral: Information
- Incentives: IMA (Experimental): Informational IMA mailer and incentive
  Interventions: Behavioral: Financial Incentives; Behavioral: Information
- Control: CDC (No Intervention): No mailer for CDC (clinical diabetes care) gap
- Information only: CDC (Experimental): Informational CDC mailer
  Interventions: Behavioral: Information
- Incentives: CDC (Experimental): Informational CDC mailer and incentive
  Interventions: Behavioral: Financial Incentives; Behavioral: Information
- Control: CCS (No Intervention): No mailer for CCS (cervical cancer screening)
- Information only: CCS (Experimental): Informational CCS mailer
  Interventions: Behavioral: Information
- Incentives: CCS (Experimental): Informational CCS mailer and incentive
  Interventions: Behavioral: Financial Incentives; Behavioral: Information
- Control: AWC (No Intervention): No mailer for AWC (adolescent well-care visit) gap
- Information only: AWC (Experimental): Informational AWC mailer
  Interventions: Behavioral: Information
- Incentives: AWC (Experimental): Informational AWC mailer and incentive
  Interventions: Behavioral: Financial Incentives; Behavioral: Information

INTERVENTIONS:
Behavioral: Financial Incentives — Incentives for gap closure.
  Arms: Incentives: AWC; Incentives: CCS; Incentives: CDC; Incentives: IMA; Incentives: LSC; Incentives: W34
Behavioral: Information — Information on care gap and closure process.
  Arms: Incentives: AWC; Incentives: CCS; Incentives: CDC; Incentives: IMA; Incentives: LSC; Incentives: W34; Information only: AWC; Information only: CCS; Information only: CDC; Information only: IMA; Information only: LSC; Information only: W34

SUMMARY:
This project seeks to understand how individuals respond to financial incentive programs for wellness care. In a randomized controlled trial among customers with care gaps, the investigators will experimentally compare the impacts of incentives for gap closure (gift cards), information on existing gaps (mailers), and no intervention. The research objectives are to assess how responsive individuals are to incentives for, and to information about, existing care gaps; and to assess spillovers from incentives onto other care. In addition, impacts on downstream utilization will be studied, which may be impacted if financial incentives are effective at increasing wellness visits.

DETAILED DESCRIPTION:
Setting and sample:

The study will be conducted among individuals enrolled in an insurance plan offered by an insurance company in the state of Nebraska.

The sample will include a subset of individuals eligible for a program designed to improve delivery of care by incentivizing individuals and their dependents to fill "care gaps" - gaps in recommended care.

Interventions:

The design will entail two overarching interventions for each incentivized care gap: Incentives, and Information Only. In addition, there will be a control that receives neither.

* Incentives. Individuals receiving the Incentives intervention for a given care gap will receive a mailer informing them of that gap, and that they are eligible for a gift card if they close that care gap.
* Information Only. Individuals receiving the Information Only intervention for a given care gap will receive a mailer informing them of that gap, but without information on the incentives available.
* Control. Individuals receiving the Control intervention for a given care gap will not receive a mailer.

All individuals will be made whole following the intervention period, regardless of treatment status; i.e. members will be compensated for closing incentivized care gaps regardless of whether they were informed of their eligibility to do so.

The specific Incentivized Care Gaps include: W34, LSC, IMA, CDC Eye Exam and/or CDC Hba1c Screening, CCS, and AWC.

Randomization:

A separate letter is sent for each care gap, so that individuals may receive more than one letter. The investigators will randomize which letters are sent.

The process will be as follows: every individual with a care gap in the sample (a care-gap, beneficiary pair) will be randomly assigned a study status: financial incentive, information only, or no letter. When it comes time to send mailers for each care gap, mailers will be sent according to the intersection of eligibility and care gap-specific treatment assignment. E.g. if at mailing time a participant is eligible for only cervical cancer screening (CCS), that participant will receive the CCS intervention (Control, Information Only, or Incentives) as pre-assigned. If the participant is also eligible for an adolescent well-visit (AWC) incentive based on her dependent's age and visit status, the participant will also receive the AWC intervention as pre-assigned; this intervention may be the same or different from her CCS intervention.

Analysis:

The investigators will compare the number and rate of care-gap closure at 6 and 18 months following the initial mailing. The investigators will also conduct heterogeneity analysis according to baseline characteristics of the population.

ELIGIBILITY:
Inclusion Criteria:

* Is a partner organization member in the region of study
* Has a care gap in one of the six target areas

Exclusion Criteria:

* Participating in another select high-intensity wellness intervention provided by the partner organization

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8042 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of care gaps closed | 6 months, from the date of randomization until end-of-year (i.e., December 31, 2018)
  Care gap closure for all care gaps. A care gap is considered closed for an individual or dependent who had not received recommended care (i.e. who had a care gap) at the time of enrollment at the time they receive the recommended care. For example, if a dependent child has not received lead screening (LSC) at the time of enrollment, the LSC care gap is considered closed once the child receives a lead screening.
Proportion of care gaps closed | 18 months, from the date of randomization until December 31, 2019
  Care gap closure for all care gaps. A care gap is considered closed for an individual or dependent who had not received recommended care (i.e. who had a care gap) at the time of enrollment at the time they receive the recommended care. For example, if a dependent child has not received lead screening (LSC) at the time of enrollment, the LSC care gap is considered closed once the child receives a lead screening.

SECONDARY OUTCOMES:
Health care expenditure during study - Total claims | 6 months, from the date of randomization until end-of-year
  (dollars)
Health care expenditure following study - Total claims | 12 months, from December 31 2018 - December 31 2019
  Total claims (dollars)
Outpatient visits during study | 6 months, from the date of randomization until end-of-year
  Number of outpatient visits
Outpatient visits following study | 12 months, from December 31 2018 - December 31 2019
  Number of outpatient visits
Inpatient visits during study | 6 months, from the date of randomization until end-of-year
  Number of inpatient visits
Inpatient visits following study | 12 months, from December 31 2018 - December 31 2019
  Number of inpatient visits
Prescriptions during study | 6 months, from the date of randomization until end-of-year
  Number of prescriptions
Prescriptions following study | 12 months, from December 31 2018 - December 31 2019
  Number of prescriptions

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided